CLINICAL TRIAL: NCT03513614
Title: Tailored Axillary Surgery With or Without Axillary Lymph Node Dissection Followed by Radiotherapy in Patients With Clinically Node-positive Breast Cancer (TAXIS). A Multicenter Randomized Phase III Trial (OPBC-03/ SAKK 23/16 /IBCSG 57-18 / ABCSG-53 / GBG-101)
Brief Title: Tailored Axillary Surgery With or Without Axillary Lymph Node Dissection Followed by Radiotherapy in Patients With Clinically Node-positive Breast Cancer (TAXIS)
Acronym: TAXIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: ETOP IBCSG Partners Foundation (Network); Austrian Breast Cancer Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-00838; ch20Weber2; 2018-000372-14 (EudraCT Number)
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Node-positive Breast Cancer
Keywords: Tailored Axillary Surgery; TAXIS; Breast Cancer; node-positive breast cancer; phase III trial; IBCSG 57-18; ABCSG
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALND (Active Comparator): Tailored axillary surgery followed by axillary lymph node dissection (ALND) and regional nodal irradiation excluding the dissected axilla.
  Interventions: Procedure: Tailored axillary surgery - both Arms; Radiation: Radiotherapy - Arm A
- No ALND (Active Comparator): Tailored axillary surgery followed by regional nodal irradiation including the full axilla.
  Interventions: Procedure: Tailored axillary surgery - both Arms; Radiation: Radiotherapy - Arm B

INTERVENTIONS:
Procedure: Tailored axillary surgery - both Arms — Axillary lymph node dissection - Arm A
Radiation: Radiotherapy - Arm A — Regional nodal irradiation excluding the dissected axilla - Arm A
  Arms: ALND
Radiation: Radiotherapy - Arm B — Regional nodal irradiation including the full axilla - Arm B
  Arms: No ALND

SUMMARY:
RATIONALE: The use of tailored axillary dissection as a tailored procedure will avoid surgical overtreatment by selectively removing the lymph nodes that are affected by the cancer, thereby sparing many women the unnecessary complications of a radical surgery, providing a better quality of life while keeping the same efficacy.

PURPOSE: The phase III trial is evaluating the optimal treatment for breast cancer patients in terms of surgery and radiotherapy.

DETAILED DESCRIPTION:
The removal of all lymph nodes in the armpit through conventional axillary dissection has been standard care for all patients with breast cancer for almost a century. In the nineties, the sentinel lymph node procedure, which involves the selective removal of the first few affected lymph nodes, was introduced in clinical practice. Today, conventional axillary dissection is still performed on many women with breast cancer that has spread to the nodes. It is the cause for relevant morbidity in the form of lymphedema, impairment of shoulder mobility, sensation disorders and chronic pain in as much as one third of all women undergoing the procedure.

The TAXIS trial will evaluate the optimal treatment for breast cancer patients in terms of surgery and radiotherapy. In particular, it will investigate the value of tailored axillary surgery (TAS), a new technique that aims at selectively removing the positive lymph nodes. TAS combines the removal of palpably suspicious nodes with the sentinel procedure. TAS is a promising procedure that may significantly decrease morbidity in breast cancer patients by avoiding surgical overtreatment.

This trial has the potential to establish a new worldwide treatment standard with hopefully less side effects and a better quality of life, while keeping the same efficacy as provided by radical surgery.

The main objective of the trial is to show that TAS and axillary radiotherapy (RT) is non-inferior to ALND in terms of disease-free survival of node positive breast cancer patients at high risk of recurrence in the era of effective systemic therapy and extended regional nodal irradiation.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria at pre-registration:

* Written informed consent according to ICH/GCP regulations prior to any trial specific procedures.
* Breast cancer, node positive detected by palpation or imaging (with or without planned neoadjuvant treatment)
* Female or male aged ≥ 18 years
* Ability to complete the Quality of Life questionnaires

Inclusion criteria at registration:

* Node-positive breast cancer (histologically or cytologically proven both in primary tumor and in lymph node) AJCC/UICC [42] stage II-III (all molecular subtypes allowed):

  * Node-positivity detected by imaging (iN+) and confirmed by pathology
  * Node-positivity detected by palpation (cN1-3) and confirmed by pathology
  * Occult breast cancer is allowed, if biopsy-proven axillary lymphatic metastasis is present
* Eligible for primary ALND or sentinel lymph node (SLN) procedure with frozen section and either:

  * Newly diagnosed
  * Isolated in-breast recurrence or second ipsilateral breast cancer after previous breast conserving surgery and sentinel procedure and at least 3 years disease free and no prior axillary dissection or axillary RT
* Most suspicious axillary lymph node clipped
* Baseline Quality of Life questionnaire has been completed
* WHO performance status 0-2
* Adequate condition for general anesthesia and breast cancer surgery
* Women with child-bearing potential are using effective contraception, are not pregnant or lactating and agree not to become pregnant during trial treatment and thereafter during the time recommended by the guidelines for adjuvant systemic therapies. A negative pregnancy test before inclusion into the trial is required for all women with child-bearing potential.
* Men agree not to father a child during trial treatment and thereafter during 6 months.

Inclusion criteria at randomization (intraoperatively)

* Node-positive breast cancer (histologically or cytologically proven both in primary tumor and in lymph node) AJCC/UICC stage II-III (all molecular subtypes allowed):

  * Node-positivity initially detected by imaging and non-palpable and residual disease confirmed by pathology** (including residual ITCs) in SLN or non SLN in case of prior neoadjuvant treatment
  * Node-positivity initially palpable and residual disease confirmed by pathology** (including residual ITCs) in case of prior neoadjuvant treatment

    * Note: patients with ypN0(i+) can be included (the AJCC stage II-III refers to the stage before neoadjuvant treatment) **Note: If the fine needle aspiration or core biopsy of the clipped node after neoadjuvant treatment unequivocally shows cancer, repeated confirmation of residual disease by intraoperative frozen section is not mandatory

Exclusion Criteria:

Exclusion criteria at pre-registration:

Any potential patient who meets any of the following criteria has to be excluded from entering the trial.

* Stage IV breast cancer
* Clinical N3c breast cancer (clinical N3a and clinical N3b are allowed)
* Clinical N2b breast cancer (clinical N2a is allowed)
* Contralateral breast cancer within 3 years Note: Contralateral Ductal Carcinoma In Situ (DCIS) is allowed if prior treatment does not interfere with or compromise the trial treatment
* Prior axillary surgery (except prior sentinel node procedure in case of in- breast recurrence)
* Prior regional radiotherapy
* History of hematologic or primary solid tumor malignancy, unless in remission for at least 3 years from pre-registration with the exception of adequately treated cervical carcinoma in situ or localized non-melanoma skin cancer.
* Treatment with any experimental drug within 30 days of pre-registration
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Exclusion criteria at randomization (intraoperatively):

Any potential patient who meets any of the following criteria has to be excluded from the trial.

* Absence of clip in the specimen radiography
* Palpable disease left behind in the axilla after Tailored Axillary Surgery (TAS)
* No SLN identified in the axilla

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2018-08-07 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2036-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | at the occurrence of the event or latest 20 years after randomization of the last patient
  The primary endpoint of this trial is DFS, defined as time from randomization until one of the following events, whichever comes first:
  * Local recurrence, regional recurrence, distant recurrence
  * Second breast cancer
  * Death from any cause Patients not experiencing an event will be censored at the date of the last available assessment.

SECONDARY OUTCOMES:
Overall survival (OS) | at the occurrence of the event or latest 20 years after randomization of the last patient
  OS will be calculated from randomization until death from any cause. Patients not experiencing an event will be censored at the last date they were known to be alive.
Breast cancer-specific survival (BCSS) | at the occurrence of the event or latest 20 years after randomization of the last patient
  BCSS will be calculated from randomization until death from breast cancer. Patients not experiencing an event will be censored at the last date they were known to be alive.
Time to local recurrence (TTLR) | at the occurrence of the event or latest 20 years after randomization of the last patient
  TTLR will be calculated from randomization until local recurrence or death from breast cancer. Patients not experiencing an event or patients who died due to other reasons before experiencing an event will be censored at the date of the last available assessment.
Time to distant recurrence (TTDR) | at the occurrence of the event or latest 20 years after randomization of the last patient
  TTDR will be calculated from randomization until distant recurrence or death from breast cancer. Patients not experiencing an event or patients who died due to other reasons before experiencing an event will be censored at the date of the last available assessment.
Physician reported morbidity outcomes (Lymphedema) | at baseline, at week 1 and 4 after surgery, before the beginning of radiotherapy. During follow-up: 9 and 12 months after randomization then every 6 months up to 3 years, then every year up to 20 years after randomization of the last patient.
Physician reported morbidity outcomes (Decreased range of shoulder motion) | at baseline, at week 1 and 4 after surgery. During follow-up: 9 and 12 months after randomization then every 6 months up to 3 years, then every year up to 10 years after randomization of the last patient.
Adverse events according to NCI CTCAE v4.03 | from date of patient consent and up to 20 years after randomization of the last patient
  Clipping-related AEs and specific AEs related to the surgical procedure and radiotherapy will be assessed according to NCI CTCAE v4.03.
Late radiotherapy-related adverse events | from date of patient consent and up to 20 years after randomization of the last patient
  Late adverse events related to the radiotherapy will be assessed according to the Late Effects in Normal Tissues-Subjective, Objective, Management and Analytic (LENT-SOMA) scale
Surgical site infections (SSI) | from date of patient consent and up to 20 years after randomization of the last patient
  SSIs will be assessed according to the Centers for Disease Control and Prevention Surgical Site Infection Classification System.

CONTACTS AND LOCATIONS:
Overall Officials: Walter P. Weber, Prof., Study Chair — University Hospital, Basel, Switzerland
Locations (67):
- United States (3):
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Duke University/Duke Cancer Center, Durham, North Carolina
  - Swedish Cancer Institute, Seattle, Washington
- Argentina (2):
  - Sanatorio Parque Breast Cancer Center, Rosario, Santa Fe Province
  - Institute of Oncology "Angel H. Roffo, Buenos Aires
- Austria (9):
  - Krankenhaus Dornbirn, Dornbirn
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Medical University of Innsbruck, Department of Gynecology, Innsbruck
  - Ordens Kinikum Linz, Barmherzige Schwestern, Linz
  - Universitätsklinik für Frauenheilkunde und Geburtshilfe; Landeskrankenhaus Salzburg der PMU, Salzburg
  - Medizinische Universität Wien - Klinik für Chirurgie, Vienna
  - Medizinische Universität Wien - Universitätsklinik für Frauenheilkunde, Vienna
  - Hanusch Hospital Vienna, Vienna
  - Klinikum Wels-Grieskrichen GmbH, Wels
- CIUSSS du Centre Ouest-de-l'Île-de-Montréal, Jewish General Hospital, Montreal, Canada
- Croatia (2):
  - Breast Centre of Clinical Hospital, Rijeka
  - HRUHC Sestre milosdrnice, Zagreb
- Germany (7):
  - Ev. Waldkrankenhaus Spandau, Berlin
  - KEM | Evang. Kliniken Essen-Mitte gGmbH, Essen
  - Niels-Stensen-Kliniken Franziskus-Hospital Harderberg, Georgsmarienhütte
  - Universitätsklinikum Heidelberg, Sektion Senologie, Heidelberg
  - ViDia Christliche Kliniken Karlsruhe, Diakonissenkrankenhaus, Karlsruhe
  - Onkologie Rheinsieg, Troisdorf
  - Helios University Hospital Wuppertal, Wuppertal
- Greece (7):
  - Attikon University Hospital, Chaïdári, Athens
  - University Hospital of Heraklion, Heraklion, Crete
  - Alexandra General Hospital, Athens
  - Larissa General University Hospital, Larissa
  - Iaso Maternity Hospital, Marousi
  - Athens Medical Center Iatriko, Marousi
  - University Hospital of Patras, Pátrai
- Hungary (3):
  - National Institute of Oncology, Budapest
  - Bacs-Kiskun Country Hospital, Kecskemét
  - University of Szeged, Szeged
- Italy (2):
  - Ospedale MultiMedica Castellanza, Castellanza
  - Fondazione Policlinico Universitario "Agostino Gemelli" di Roma, Rome
- Pauls Stradinš Clinical University Hospital, Riga, Latvia
- National Cancer Institut, Vilnius, Lithuania
- South Korea (2):
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
- Switzerland (27):
  - Kantonsspital Aarau, Aarau
  - Brustzentrum Basel und Netzwerk, Allschwil
  - Kantonsspital Baden, Baden
  - Universitätsspital Basel, Basel
  - Bethesda Spital Basel, Gynäkologie und Geburtshilfe, Basel
  - St. Claraspital AG, Basel
  - Brustzentrum Bern, Lindenhofgruppe Centerclinic, Bern
  - Clinique de Grangettes, Chêne-Bougeries
  - Kantonsspital Graubünden, Chur
  - Brustzentrum Thurgau, Frauenfeld
  - Breast center Fribourg, Fribourg
  - HUG - Hôpitaux Universitaires de Genève, Geneva
  - Clinique de Genolier, Genolier
  - Hôpital Neuchâtelois, La Chaux-de-Fonds
  - Centre Hospitalier Universitaire Vaudois CHUV, Lausanne
  - Luzerner Kantonsspital - Brustzentrum, Lucerne
  - Hirslanden Klinik St. Anna, Lucerne
  - Centro di Senologia della Svizzera Italiana CSSI, Lugano
  - Kantonsspital St. Gallen, Sankt Gallen
  - Tumor-and Breast centre Ostschweiz, Sankt Gallen
  - Spital Limmattal, Schlieren
  - Hôpital du Valais / Hôpital de Sion, Sion
  - Kantonsspital Winterthur, Brustzentrum, Winterthur
  - Spital Zollikerberg, Zollikerberg
  - Brust-Zentrum Zürich (Seefeld), Zurich
  - Stadtspital Triemli, Zurich
  - Universitäts Spital Zürich, Zurich

REFERENCES:
- [Result] Weber WP, Matrai Z, Hayoz S, Tausch C, Henke G, Zwahlen DR, Gruber G, Zimmermann F, Seiler S, Maddox C, Ruhstaller T, Muenst S, Ackerknecht M, Kuemmel S, Bjelic-Radisic V, Kurzeder C, Ujhelyi M, Vrieling C, Satler R, Meyer I, Becciolini C, Bucher S, Simonson C, Fehr PM, Gabriel N, Maraz R, Sarlos D, Dedes KJ, Leo C, Berclaz G, Dubsky P, Exner R, Fansa H, Hager C, Reisenberger K, Singer CF, Reitsamer R, Reinisch M, Winkler J, Lam GT, Fehr MK, Naydina T, Kohlik M, Clerc K, Ostapenko V, Fitzal F, Nussbaumer R, Maggi N, Schulz A, Markellou P, Lelievre L, Egle D, Heil J, Knauer M. Tailored axillary surgery in patients with clinically node-positive breast cancer: Pre-planned feasibility substudy of TAXIS (OPBC-03, SAKK 23/16, IBCSG 57-18, ABCSG-53, GBG 101). Breast. 2021 Dec;60:98-110. doi: 10.1016/j.breast.2021.09.004. Epub 2021 Sep 8. PMID 34555676
- [Derived] Weber WP, Heidinger M, Hayoz S, Matrai Z, Tausch C, Henke G, Zwahlen DR, Gruber G, Zimmermann F, Montagna G, Andreozzi M, Goldschmidt M, Schulz A, Mueller A, Ackerknecht M, Tampaki EC, Bjelic-Radisic V, Kurzeder C, Savolt A, Smanyko V, Hagen D, Muller DJ, Gnant M, Loibl S, Fitzal F, Markellou P, Bekes I, Egle D, Heil J, Knauer M. Impact of Imaging-Guided Localization on Performance of Tailored Axillary Surgery in Patients with Clinically Node-Positive Breast Cancer: Prospective Cohort Study Within TAXIS (OPBC-03, SAKK 23/16, IBCSG 57-18, ABCSG-53, GBG 101). Ann Surg Oncol. 2024 Jan;31(1):344-355. doi: 10.1245/s10434-023-14404-4. Epub 2023 Oct 30. PMID 37903951
- [Derived] Tausch C, Daster K, Hayoz S, Matrai Z, Fitzal F, Henke G, Zwahlen DR, Gruber G, Zimmermann F, Andreozzi M, Goldschmidt M, Schulz A, Maggi N, Saccilotto R, Heidinger M, Mueller A, Tampaki EC, Bjelic-Radisic V, Savolt A, Smanyko V, Hagen D, Muller DJ, Gnant M, Loibl S, Markellou P, Bekes I, Egle D, Ruhstaller T, Muenst S, Kuemmel S, Vrieling C, Satler R, Becciolini C, Bucher S, Kurzeder C, Simonson C, Fehr PM, Gabriel N, Maraz R, Sarlos D, Dedes KJ, Leo C, Berclaz G, Fansa H, Hager C, Reisenberger K, Singer CF, Montagna G, Reitsamer R, Winkler J, Lam GT, Fehr MK, Naydina T, Kohlik M, Clerc K, Ostapenko V, Lelievre L, Heil J, Knauer M, Weber WP. Trends in use of neoadjuvant systemic therapy in patients with clinically node-positive breast cancer in Europe: prospective TAXIS study (OPBC-03, SAKK 23/16, IBCSG 57-18, ABCSG-53, GBG 101). Breast Cancer Res Treat. 2023 Sep;201(2):215-225. doi: 10.1007/s10549-023-06999-9. Epub 2023 Jun 25. PMID 37355526
- [Derived] Henke G, Knauer M, Ribi K, Hayoz S, Gerard MA, Ruhstaller T, Zwahlen DR, Muenst S, Ackerknecht M, Hawle H, Fitzal F, Gnant M, Matrai Z, Ballardini B, Gyr A, Kurzeder C, Weber WP. Tailored axillary surgery with or without axillary lymph node dissection followed by radiotherapy in patients with clinically node-positive breast cancer (TAXIS): study protocol for a multicenter, randomized phase-III trial. Trials. 2018 Dec 4;19(1):667. doi: 10.1186/s13063-018-3021-9. PMID 30514362

DOCUMENTS (1):
  • Informed Consent Form (2024-01-11): https://cdn.clinicaltrials.gov/large-docs/14/NCT03513614/ICF_000.pdf